CLINICAL TRIAL: NCT00339599
Title: Study of Chemokine Markers and Genes as Predictors of Cardiovascular Disease
Brief Title: Genetic Predictors of Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905247; 05-C-N247
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2015-08-03

CONDITIONS: Cardiovascular Disease
Keywords: Atherosclerosis; Single Nucleotide Polymorphisms; Monocyte Chemotactic Protein-1; Inflammation; Eotaxin
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Inflammation

SUMMARY:
This study, conducted in collaboration with the Johns Hopkins University School of Medicine, will explore the genetic influences on susceptibility to atherosclerotic cardiovascular disease (ASCVD). Atherosclerosis is a chronic narrowing of the arteries caused by an incremental buildup of fatty substances on the linings of walls of arteries. This study will examine the role of genes related to the inflammatory process on the incidence of ASCVD and on levels of chemokines (proteins involved in inflammation).

DNA samples, chemokines levels and relevant clinical data from patients enrolled in Johns Hopkins's sibling and family heart studies are analyzed for specific gene markers. The studies include: Nurse Model in Black Families at Risk for Heart Disease; Genotypic Determinants of Aspirin Response in High Risk Families; and Coronary Disease Detection by Thallium SPECT and Fast CT. All of the enrolled patients have consented to have their DNA used for testing of genetic factors that may predict cardiovascular disease and do not contain patient identifier information.

DETAILED DESCRIPTION:
Background:

Atherosclerosis is a chronic inflammatory disease classically triggered by hypertension, diabetes, smoking and elevated cholesterol.

It is hypothesized that genetic predisposition plays a crucial role in an individual's susceptibility to these risk factors with Single Nucleotide Polymorphisms (SNPs) being identified as functional mediators of key inflammatory genes.

Objectives:

To determine the frequency of haplotypes of SNP combinations in the proximal promoter region of MCP-1, the MCP-3 gene, and eotaxin gene in patients with risk factors for CVD and their siblings.

To determine the MCP-1 levels in an affected population with Coronary artery disease and their siblings and certain haplotypes to determine a functional association between MCP-1 levels and haplotype frequency.

Eligibility:

Eligibility criteria for enrollment in sib and family studies included: 1) having a sib or 1st degree family member with heart disease, 2) ability to give inform consent to participate in the study, 3) age 18 years or older, 4) ability to speak English or Spanish. The entire set of 2,000 samples available to the LDG will be analyzed. No subject will be excluded.

Design:

DNAs derived from properly consented subjects enrolled in three protocols sponsored by the Johns Hopkins Heart Study will be sent to the LGD and used to test specific markers in the MCP-1, MCP-3, and eotaxin chemokine family located in the C-C chemokine cluster on chromosome17q11.2.

A minimum of 11 SNPs will be examined.

Sib-pair analysis will be utilized to identify associated markers. Linear regressions will be used to analyze associations between genetic variations and chemokine levels. Haplotype will be assigned to unrelated individuals using the maximum likelihood approach.

The DNA samples, chemokine levels, and relevant clinical data provided by John Hopkins University School of Medicine will be coded and linked.

Following this study, the DNAs will be maintained in our repository and curated through our central Laboratory database. Loss or destruction of these samples will be annotated to our database and cannot impact the study participants in any way. We understand that studies subsequent to the completion of this protocol will require additional OHSR/IRB approval prior to commencement.

ELIGIBILITY:
* INCLUSION CRITERIA

Have a sibling or first degree family member with heart disease

Ability to give informed consent to participate in the study

Age 18 years or older

Ability to speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2306 (Actual)
Dates: Start 2005-09-20; Study Completion 2015-08-03

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Cortner, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Francis SE, Camp NJ, Dewberry RM, Gunn J, Syrris P, Carter ND, Jeffery S, Kaski JC, Cumberland DC, Duff GW, Crossman DC. Interleukin-1 receptor antagonist gene polymorphism and coronary artery disease. Circulation. 1999 Feb 23;99(7):861-6. doi: 10.1161/01.cir.99.7.861. PMID 10027806
- [Background] Rovin BH, Lu L, Saxena R. A novel polymorphism in the MCP-1 gene regulatory region that influences MCP-1 expression. Biochem Biophys Res Commun. 1999 Jun 7;259(2):344-8. doi: 10.1006/bbrc.1999.0796. PMID 10362511